CLINICAL TRIAL: NCT03350789
Title: Efficacy and Mechanism of Acupuncture on Patients With Chronic Sciatica Using fMRI: A Randomized, Patient-Assessor Blind, Sham-Controlled Clinical Trial
Brief Title: Efficacy and Mechanism of Acupuncture for Chronic Sciatica Using fMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Mi-Yeon Song, Professor, K.M.D., Ph.D., Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KHNMC OH 2017-08-004-002
Record Dates: First submitted 2017-11-15; First posted 2017-11-22 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Chronic Sciatica
Keywords: acupuncture; sciatica; MRI, functional
MeSH Terms: conditions — Sciatica

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real acupuncture (Experimental): manual acupuncture + electroacupuncuture on acupoints, twice a week, for 4 weeks
  Interventions: Device: Real acupuncture
- Sham acupuncture (Sham Comparator): sham acupuncture (no skin penetration) + placebo electroacupuncture without electrical stimulation on acupoints, twice a week, for 4 weeks
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Real acupuncture — manual acupuncture(0.25mm diameter x 40mm length, stainless steel, Dongbangacupuncture Inc., Korea) (unilateral GB30) + electroacupuncture(0.25mm diameter x 40mm length, stainless steel, Dongbangacupuncture Inc., Korea) (unilateral EX-B2 (L4 & L5), BL25, BL23, BL40, GB34), twice a week, for 4 weeks, common approaches for the treatment of chronic sciatica used by doctors of Korean medicine in Korea today
  Arms: Real acupuncture
Device: Sham acupuncture — sham acupuncture without skin penetration(0.25mm diameter x 40mm length, stainless steel, Acuprime, UK) (unilateral GB30) + placebo electroacupuncture (0.25mm diameter x 40mm length, stainless steel, Dongbangacupuncture Inc., Korea) without electrical stimulation (unilateral EX-B2, BL25, BL23, BL40, GB34), twice a week, for 4 weeks
  Arms: Sham acupuncture

SUMMARY:
This research is planned to build a basis about the efficacy and mechanism of acupuncture on pain and emotional disorder in patients with chronic sciatica using fMRI.

DETAILED DESCRIPTION:
Clinical research to assess the effect of acupuncture for chronic sciatica on pain and emotional disorder will be processed with randomized, patient-assessor blinding, and sham-acupuncture controlled study design. Sixty eight subjects would be collected and divided into two groups(experimental and placebo, 34 subjects each). Experimental group will undergo with real acupuncture treatment(manual acupuncture + electroacupuncture) and placebo group will undergo with sham acupuncture treatment (acupuncture without skin penetration + electroacupuncture without electrical stimulation) twice a week, for 4 weeks. The effect on parameters related with pain and emotional disorder will be assessed at 1(baseline: just before the beginning of treatment) and 5(primary end point: 1 week after the end of treatment) weeks. Functional magnetic resonance imaging will be also conducted for 52 subjects(experimental and placebo, 20 among 34 subjects each + normal control 12 subjects) at 1 and 5 weeks to seek machanism of acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* adults 19 years of age or more and 70 years of age or less
* clinical diagnosis of chronic sciatica (pain lasting 3 months or more)
* 40mm or more of 100mm VAS for bothersomeness due to sciatica
* volunteers through announcements and advertisements with written informed consent

Exclusion Criteria:

* spinal surgery within the past 6 months
* diagnosis of specific severe diseases resulting in sciatica: malignant tumor, spinal infection, inflammatory sponlylitis
* progressive neurological deficit or severe neurological signs
* other chronic diseases which could disturb the effect of treatments and the results of the study: cardiovascular diseases, autoimmune diseases, renal diseases, diabetic neuropathy, dementia, epilepsy
* inadequate or insafe for the treatment of acupuncture/ electroacupuncture: hemorrhagic diseases, medication of anticoagulant, serious diabetes mellitus vulnerable to infections, serious cardiovascular diseases/ pacemaker, metal materials interior of the body
* currently or might be pregnant
* severe mental illness
* currently participating other clinical trials
* experience of acupuncture or electroacupuncture treatment, or taking medicines which might affect the symptom of pain such as corticosteroids, narcotics, NSAIDs or considered to be inadequate by the investigators within the past week (But they could be included only after going through 2 weeks of wash out period.)
* difficulty of writing informed consent
* inadeguate or insafe for MRI scanning: claustrophobia, metal materials interor of the body
* other inadequate subjects assessed by the study investigators

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale for bothersomeness | baseline, 1-1, 1-2, 2-1, 2-2, 3-1, 3-2, 4-1, 4-2, 5, and 8 weeks
  change in visual analoge scale for bothersomeness [range: 0(better)-100(worse) mm]

SECONDARY OUTCOMES:
Visual analogue scale for pain intensity | baseline, 1-1, 1-2, 2-1, 2-2, 3-1, 3-2, 4-1, 4-2, 5, and 8 weeks
  change in visual analogue scale for pain intensity [range: 0(better)-100(worse) mm]
Oswestry Disability Index | week 1(before treatment) and week 5(1 week after treatment, primary endpoint)
  change in functional scale: Oswestry Disability Index [10 items, 0-5 points each, total 0(better) -50(worse) points]
EuroQol 5-Dimension | week 1(before treatment) and week 5(1 week after treatment, primary endpoint)
  change in quality of life scale: EuroQol 5-Dimension [5 items, 1-3 points each, total 5(better) -15(worse) points]
Coping Strategy Questionnaire | week 1(before treatment) and week 5(1 week after treatment, primary endpoint)
  change in coping scale: Coping Strategy Questionnaire [8 subscales, total 48 items, 0-6 points each, divided into adaptive coping or disadaptive coping, not better or worse]
Beck Depression Inventory | week 1(before treatment) and week 5(1 week after treatment, primary endpoint)
  change in emotion scale: Beck Depression Inventory [21 items, 1-4 points each, total 21(better) -84(worse) points]
State-Trait Anxiety Inventory | week 1(before treatment) and week 5(1 week after treatment, primary endpoint)
  change in emotion scale: State-Trait Anxiety Inventory [40 items, 1-4 points each, divided into state anxiety or trait anxiety, not better or worse]
blood oxygenation level dependent in Magnetic Resonance Image, functional | week 1(before treatment) and week 5(1 week after treatment, primary endpoint)
  change in blood oxygenation level dependent of steady state and event-related block design scan run in functional magnetic resonance image.
  cf. functional magnetic resonance image scan run design: REST(6 min)-TASK1(5 min)-3D T1(5 min)-TASK2(5 min)-DTI(6 min)-TASK3(6 min).
  REST: steady-state resting scan run. TASK1/2: event-related block design, emotion and pain stimulation model scan run. 2 distinct 5-min experiment blocks (each block-20(5*4) stimuli (6 sec, inter-stimulus interval: 9 sec); comprised of visual picture(International Affective Picture System: neutral, negative), pain(low back, hand), picture plus pain).
  3D T1: structural image acquisition. DTI: diffusion tensor imaging. TASK3: steady state pain model scan run. Low back extension pain model.
Adverse events | baseline, 1-1, 1-2, 2-1, 2-2, 3-1, 3-2, 4-1, 4-2, 5, and 8 weeks
  number of participants with adverse events
  * assessment of severity: mild, moderate, severe
  * assessment of relation: definitely related, probably related, possibly related, probably not related, definitely not related, unknown

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Yeon Song, Ph.D., Principal Investigator — Department of Rehabilitation Medicine of Korean Medicine, Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim KW, Park K, Park HJ, Jahng GH, Jo DJ, Cho JH, Song EM, Shin WC, Yoon YJ, Kim SJ, Eun S, Song MY. Effect and neurophysiological mechanism of acupuncture in patients with chronic sciatica: protocol for a randomized, patient-assessor blind, sham-controlled clinical trial. Trials. 2019 Jan 16;20(1):56. doi: 10.1186/s13063-018-3164-8. PMID 30651139